CLINICAL TRIAL: NCT01879683
Title: A Phase 1b, Multicenter, Open Label Study Evaluating Safety, Tolerability and Preliminary Efficacy of LiRIS® 400 mg in Women With Ulcerative Interstitial Cystitis
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of LiRIS® 400 mg in Women With Interstitial Cystitis (IC) and Hunner's Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: TARIS Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAR-100-105
Record Dates: First submitted 2013-06-10; First posted 2013-06-18 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Interstitial Cystitis
Keywords: Hunner's lesion
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LiRIS® 400 mg (Experimental): LiRIS® 400 mg (Lidocaine Releasing Intravesical System 400 mg); a drug-device combination product, placed in the urinary bladder, and releases lidocaine into the bladder over a 14 day period.
  Interventions: Drug: LiRIS® 400 mg

INTERVENTIONS:
Drug: LiRIS® 400 mg — LiRIS® 400 mg is a drug-device combination product which is placed in the bladder during cystoscopy, remains in the bladder for up to 14 days gradually releasing lidocaine, and removed from the bladder via cystoscopy.

SUMMARY:
The purpose of the study is to evaluate if LiRIS 400 mg is safe and tolerable when administered to women with Interstitial Cystitis with Hunner's lesions, and to evaluate any change in the bladder or in IC symptoms, following LiRIS administration.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 and older
* Interstitial Cystitis with history of Hunner's lesions in the bladder
* Moderate to severe bladder discomfort
* Confirmation of Hunner's lesions in Bladder
* Able to report symptom (pain and voiding frequency) in a diary throughout the study

Exclusion Criteria:

* Pregnant women
* History or presence of bladder cancer
* History or presence of any condition that would make it difficult to evaluate bladder symptoms

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Corewell Health East
Locations (2):
- United States (2):
  - Advance Urology Institute, Daytona Beach, Florida
  - William Beaumont Hospital, Royal Oak, Michigan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LiRIS® 400 mg
Started | 10
Completed | 9
Not Completed | 1
Not completed — Did not Complete 4-week Follow-up Visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | LiRIS® 400 mg
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants by Change From Baseline in Appearance of Hunner's Lesions at Day 14
Description: The appearance of the Hunner's lesions was assessed by the investigator using video capture of the bladder mucosa during the cystoscopic examinations. Complete responders (CR)=no lesions observed at day of last LiRIS removal; Partial responders (PR)=presence of residual lesions on day of last LiRIS removal however there is cystoscopic evidence of a decrease in either: i) the affected area as calculated by size and dimension of individual lesions summed together or ii) the lesion number or iii) the lesion(s) severity (mild, moderate, severe) as compared with Baseline assessment; Stable Disease=no change in the appearance of lesions and no new lesions on day of last LiRIS removal compared with Baseline assessment; Non-responders=worsening of mucosal appearance on day of last LiRIS removal.
Time Frame: Baseline, Day 14
Population: Per protocol population included all participants who retained each LiRIS for both 14-day treatment periods and then completed the 4-week follow-up visit without any major protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | LiRIS® 400 mg
Number analyzed (Participants) | 7
percentage of participants
  Complete Responders | 0.0
  Partial Responders | 85.7
  Stable Disease | 14.3
  Non-Responders | 0.0

2. Secondary Outcome: Change From Baseline in Patient Reported Interstitial Cystitis (IC) Symptom: Average Bladder Pain
Description: Participants rated symptom bladder pain averaged over the previous 3 days using an 11-point numeric rating scale where: 0=no pain to 10=worst pain imaginable. A negative change from Baseline indicates improvement.
Time Frame: Baseline, during treatment (Days 7, 14, 20, 28) and during follow up (Weeks 1, 2, 4, 8, 12)
Population: Per protocol population included all participants who retained each LiRIS for both 14-day treatment periods and then completed the 4-week follow-up visit without any major protocol deviations. 2 participants did not have data at Week 8 and 12 Follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | LiRIS® 400 mg
Number analyzed (Participants) | 7
score on a scale
  Baseline | 5.46 (1.955)
  Change from Baseline at Day 7 | -1.71 (1.494)
  Change from Baseline at Day 14 | -2.97 (1.739)
  Change from Baseline at Day 20 | -4.00 (2.498)
  Change from Baseline at Day 28 | -4.27 (2.411)
  Change from Baseline at Week 1 Follow-up | -4.11 (2.753)
  Change from Baseline at Week 2 Follow-up | -3.70 (2.922)
  Change from Baseline at Week 4 Follow-up | -3.69 (2.781)
  Change from Baseline at Week 8 Follow-up (n=5) | -3.72 (3.371)
  Change from Baseline at Week 12 Follow-up (n=5) | -4.40 (2.939)

3. Secondary Outcome: Change From Baseline in Patient Reported IC Symptom: Daily Total Voids
Description: The number of day-time voidings and the number of night-time voidings were averaged over a period of 3 full days and nights. A negative change from Baseline indicates improvement
Time Frame: Baseline, during treatment (Days 7, 14, 20, 28) and during follow-up (Weeks 1, 2, 4, 8, 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: voids
Arm/Group | LiRIS® 400 mg
Number analyzed (Participants) | 7
voids
  Baseline | 18.2 (5.74)
  Change from Baseline at Day 7 | -3.3 (2.27)
  Change from Baseline at Day 14 | -3.5 (3.95)
  Change from Baseline at Day 20 | -5.7 (2.18)
  Change from Baseline at Day 28 | -5.5 (2.46)
  Change from Baseline at Week 1 Follow-up | -5.3 (3.67)
  Change from Baseline at Week 2 Follow-up | -4.5 (4.41)
  Change from Baseline at Week 4 Follow-up | -5.4 (4.29)
  Change from Baseline at Week 8 Follow-up (n=5) | -4.9 (4.42)
  Change from Baseline at Week 1 Follow-up (n=5) | -3.9 (4.42)

4. Primary Outcome: Percentage of Participants by Change From Baseline in Appearance of Hunner's Lesions at Day 28
Description: The appearance of the Hunner's lesions was assessed by the investigator using video capture of the bladder mucosa during the cystoscopic examinations. Complete responders (CR)=no lesions observed at day of last LiRIS removal; Partial responders (PR) = presence of residual lesions on day of last LiRIS removal however there is cystoscopic evidence of a decrease in either i) the affected area as calculated by size and dimension of individual lesions summed together or ii) the lesion number or iii) the lesion(s) severity (mild, moderate, severe) as compared with Baseline assessment; Stable Disease=no change in the appearance of lesions and no new lesions on day of last LiRIS removal compared with Baseline assessment; Non-responders=worsening of mucosal appearance on day of last LiRIS removal.
Time Frame: Baseline, Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | LiRIS® 400 mg
Number analyzed (Participants) | 7
percentage of participants
  Complete Responders | 0.0
  Partial Responders | 100.0
  Stable Disease | 0.0
  Non-Responders | 0.0

ADVERSE EVENTS:
Arm/Group | LiRIS® 400 mg
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 6/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LiRIS® 400 mg (N=10)
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Proctalgia (Gastrointestinal disorders) | 1
Cystitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral swelling (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Blood urine present (Investigations) | 1
White blood cells urine positive (Investigations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.